CLINICAL TRIAL: NCT07103330
Title: Evaluation of Cranial Flap Fixation With Montage Flowable Settable Bone Paste
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abyrx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Abyrx PMRCT 25-001
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Cranial Bone; Post-operative Complications; Cranial Fixation; Cranioplasty; Adhesive Bone Cement
Keywords: Cranioplasty; Settable bone paste; Adhesive cranial cement

STUDY DESIGN:
Intervention Model Description: Post-market, Prospective, Randomized, Multi Center, Single Blind (Patient)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Montage Flowable Settable Bone Paste (Experimental): Fixation using Montage Flowable Settable Bone Paste exclusively
  Interventions: Device: Cranial flap placement and fixation using only Montage Flowable Settable Bone Paste
- Control (Active Comparator): Metallic fixation hardware
  Interventions: Device: Metallic fixation hardware

INTERVENTIONS:
Device: Metallic fixation hardware — Control
  Arms: Control
Device: Cranial flap placement and fixation using only Montage Flowable Settable Bone Paste — Experimental
  Arms: Montage Flowable Settable Bone Paste

SUMMARY:
Montage Flowable Settable Bone Paste is a self-setting calcium phosphate cement indicated for use in the repair of neurosurgical burr holes, contiguous craniotomy cuts and other cranial defects with a surface area no larger than 25cm2. It is also intended to be used for the fixation of cranial bone flaps following craniotomy. The MONTAGE Flowable device comprises two separate components of paste-like consistency containing granular calcium phosphate, calcium stearate, vitamin E acetate, a triglyceride, polyalcohols and a mixture of a lactide-diester and polyester-based polymers. When mixed together in the applicator tip, the components of the MONTAGE Flowable device form a cohesive paste-like material that adheres to the bone surface and remains in place following application. The resulting hardened, resorbable material is primarily calcium phosphate. The components must be mixed immediately prior to use.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 years of age
2. Undergoing a cranial procedure in supratentorial location
3. Width of craniotomy kerf line <3mm for than 75% of the bone flap border

Exclusion Criteria:

1. Subject requires a procedure involving a translabyrinthine, transsphenoidal, transoral approach, or any procedure that penetrates the air sinus or mastoid air cells.
2. Subject has clinically significant hydrocephalus or clinical evidence of altered CSF dynamics.
3. Subject has undergone a previous, open intracranial neurosurgical procedure in the same anatomical location. (Note: stereotactic biopsy was not exclusionary).
4. Subject requires a craniectomy (the bone flap is not replaced during the current surgery).
5. Subject had radiation treatment to the surgical site, or standard fractionated radiation therapy was planned post index-procedure. (Note: stereotactic radiosurgery prior to the planned index procedure was not an exclusion criterion.)
6. Subject requires a craniotomy across the sinus for which Montage Flowable is applied adjacent to or within the sinus to fixate the cranial flap.
7. Subject has a condition with anticipated survival shorter than six months.
8. Subject has undergone chemotherapy treatment, excluding hormonal therapy, within three weeks prior to the planned index procedure, or use of intracavitary chemotherapy wafer (BCNU) was planned, or chemotherapy treatment was planned within two weeks after the index procedure was performed.
9. Standard use of peri-operative steroids (i.e., corticosteroids) is permitted. Chronic steroid use (defined as daily use of corticosteroids for ≥ 8 weeks) for the purposes of reducing the side effects of chemotherapy and/or radiation therapy for cancer is not exclusionary unless the patient is deemed by the investigator to be suffering from steroid toxicity (i.e., Cushing's syndrome) manifested by symptoms and signs such as thin skin, striae, easy bruising, muscle atrophy, upper body obesity, severe fatigue, etc. Use of corticosteroids on a chronic basis (as defined previously) for purposes other than decreasing the symptoms of systemic chemotherapy is exclusionary unless those steroids were discontinued 4 weeks prior to the planned index procedure.
10. Subject receives warfarin, heparin, other anticoagulant agents on a daily basis and pre-surgical, standard of care drug wash-out did not occur.
11. Subject is pregnant, breast-feeding, or intended to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cranial flap immobility | 12 months
  Cranial flap immobility as determine by the neurosurgeon will be tabulated and compared between group

SECONDARY OUTCOMES:
Flap localization | 12 months
  Localization of the flap based on CT scan compared between groups.
Device-related adverse events | 12 months
  • Device related adverse events included all adverse events classified as definitely, probably, possibly, or undetermined relation to the device or procedure

OTHER OUTCOMES:
Complications | 12 months
  Complication categories will also be tabulated and compared

IPD SHARING:
Plan to Share IPD: No